CLINICAL TRIAL: NCT00000565
Title: Clinical Study of Intermittent Positive Pressure Breathing (IPPB)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: 203
Record Dates: First submitted 1999-10-27; First posted 1999-10-28 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2002-05

CONDITIONS: Lung Diseases; Lung Diseases, Obstructive; Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Lung Diseases; Lung Diseases, Obstructive; Pulmonary Disease, Chronic Obstructive | interventions — Intermittent Positive-Pressure Breathing

INTERVENTIONS:
Procedure: intermittent positive-pressure breathing

SUMMARY:
To evaluate the efficacy of long-term intermittent positive pressure breathing (IPPB) treatment when used as an adjunct to the overall care of ambulatory outpatients with chronic obstructive pulmonary disease. The evaluation compared the use of IPPB with use of a powered nebulizer.

DETAILED DESCRIPTION:
BACKGROUND:

Intermittent positive pressure breathing may be a useful adjunct therapy for patients with chronic obstructive pulmonary disease. It is, however, quite expensive; moreover, in 1976 its treatment efficacy had not been determined. Although the effectiveness of IPPB had been previously studied, the influence of long-term treatment was not known for the following reasons: The individuals studied had been too few and were not randomly assigned to treatment groups, the patient groups were not homogeneous and their clinical and functional status were not well-documented, and precise descriptions of the manner in which IPPB was administered were not recorded.

Based on these facts, a conference on the Scientific Basis of Respiratory Therapy, co-sponsored by the American Thoracic Society and the Division of Lung Diseases, issued a recommendation to develop a controlled clinical study of IPPB. Contracts were awarded to five clinical centers and a data center in November 1976. Planning of the trial ended in November 1977. Recruitment began in April 1978 for the 985 individuals who took part in this trial and ended in October 1980. Patients enrolled after March 31, 1980, were followed for 30 months instead of 36 months. Follow-up was completed in May 1983.

DESIGN NARRATIVE:

Randomized, fixed sample of 985 patients. Eligible patients were assigned to a treatment group using intermittent positive pressure breathing or to a control group using a powered nebulizer for treatment 3-4 times a day. Treatments continued for 3 years. Endpoints related to quality of life and respiratory function and capability.

ELIGIBILITY:
Men and women, ages 30 to 74, who were ambulatory and had symptomatic chronic bronchitis or emphysema.

Ages: 30 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1976-11

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Anthonisen — University of Manitoba; John Hodgkin — Loma Linda University Medical Center; Philip Hopewell — San Francisco General Hospital; David Levin — University of Oklahoma; Paul Stevens — Baylor College of Medicine; Elizabeth Wright — George Washington University

REFERENCES:
- [Background] National Heart, Lung, and Blood Institute, Division of Lung Diseases: Protocol for Intermittent Positive Pressure Breathing Collaborative Program. Bethesda, Maryland: National Institutes of Health, 1978.
- [Background] Hodgkin JE and Zorn EG: Intermittent Positive Pressure Breathing (IPPB) in the Outpatient Management of Chronic Obstructive Pulmonary Disease (COPD): Description of the NIH Clinical Trial. Respiratory Care, 26:1095-1104, 1981.
- [Background] Intermittent positive pressure breathing therapy of chronic obstructive pulmonary disease. A clinical trial. Ann Intern Med. 1983 Nov;99(5):612-20. doi: 10.7326/0003-4819-99-5-612. PMID 6357018
- [Background] Prigatano GP, Parsons O, Wright E, Levin DC, Hawryluk G. Neuropsychological test performance in mildly hypoxemic patients with chronic obstructive pulmonary disease. J Consult Clin Psychol. 1983 Feb;51(1):108-16. doi: 10.1037//0022-006x.51.1.108. No abstract available. PMID 6826857
- [Background] Prigatano GP, Wright EC, Levin D. Quality of life and its predictors in patients with mild hypoxemia and chronic obstructive pulmonary disease. Arch Intern Med. 1984 Aug;144(8):1613-9. PMID 6380440
- [Background] Nagai A, West WW, Paul JL, Thurlbeck WM. The National Institutes of Health Intermittent Positive-Pressure Breathing trial: pathology studies. I. Interrelationship between morphologic lesions. Am Rev Respir Dis. 1985 Nov;132(5):937-45. doi: 10.1164/arrd.1985.132.5.937. PMID 3904548
- [Background] Nagai A, West WW, Thurlbeck WM. The National Institutes of Health Intermittent Positive-Pressure Breathing trial: pathology studies. II. Correlation between morphologic findings, clinical findings, and evidence of expiratory air-flow obstruction. Am Rev Respir Dis. 1985 Nov;132(5):946-53. doi: 10.1164/arrd.1985.132.5.946. PMID 3904549
- [Background] West WW, Nagai A, Hodgkin JE, Thurlbeck WM. The National Institutes of Health Intermittent Positive Pressure Breathing trial--pathology studies. III. The diagnosis of emphysema. Am Rev Respir Dis. 1987 Jan;135(1):123-9. doi: 10.1164/arrd.1987.135.1.123. PMID 3541712
- [Background] Wilson DO, Rogers RM, Wright EC, Anthonisen NR. Body weight in chronic obstructive pulmonary disease. The National Institutes of Health Intermittent Positive-Pressure Breathing Trial. Am Rev Respir Dis. 1989 Jun;139(6):1435-8. doi: 10.1164/ajrccm/139.6.1435. PMID 2658702
- [Background] Matsuba K, Ikeda T, Nagai A, Thurlbeck WM. The National Institutes of Health Intermittent Positive-Pressure Breathing Trial: pathology studies. IV. The Destructive index. Am Rev Respir Dis. 1989 Jun;139(6):1439-45. doi: 10.1164/ajrccm/139.6.1439. PMID 2658703
- [Background] Intermittent Positive Pressure Breathing Trial Group. (Letter). Ann Intern Med, 100:458, 1984.
- Available data/document: Individual Participant Data Set: IPPB — http://biolincc.nhlbi.nih.gov/studies/ippb/ — NHLBI provides controlled access to IPD through BioLINCC. Access requires registration, evidence of local IRB approval or certification of exemption from IRB review, and completion of a data use agreement.
- Available data/document: Study Protocol — http://biolincc.nhlbi.nih.gov/studies/ippb/
- Available data/document: Study Forms — http://biolincc.nhlbi.nih.gov/studies/ippb/
- Available data/document: Manual of Procedures — http://biolincc.nhlbi.nih.gov/studies/ippb/